CLINICAL TRIAL: NCT05414149
Title: Efficacy and Safety Comparison of Ranibizumab and Conbercept Pretreatment Before Vitrectomy in Proliferative Diabetic Retinopathy
Brief Title: Efficacy and Safety Comparison of IVR and IVC Before Vitrectomy in Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PKUPHophthalmol
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy; ranibizumab; conbercept
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVR group (Active Comparator): Patients that received intravitreal ranibizumab injections (IVR) (0.5mg/0.05ml) before vitreous surgery were assigned to IVR group 3-5 days before three-port transconjunctival 25-G pars plana vitrectomy (PPV). All patients underwent 25-gauge transconjunctival sutureless vitrectomy using the 25-gauge Constellation system (Alcon, Fort Worth, TX, USA) system under local or anesthesia. A speed of 5000 cuts per minute was used for vitrectomy.
  Interventions: Procedure: preoperative intravitreal injections of ranibizumab or conbercept
- IVC group (Experimental): Patients that received intravitreal conbercept injection (IVC) (0.5mg/0.05ml) before vitreous surgery were assigned to IVC group 3-5 days before three-port transconjunctival 25-G pars plana vitrectomy (PPV). All patients underwent 25-gauge transconjunctival sutureless vitrectomy using the 25-gauge Constellation system (Alcon, Fort Worth, TX, USA) system under local or anesthesia. A speed of 5000 cuts per minute was used for vitrectomy.
  Interventions: Procedure: preoperative intravitreal injections of ranibizumab or conbercept

INTERVENTIONS:
Procedure: preoperative intravitreal injections of ranibizumab or conbercept — IVR group means patients received intravitreal ranibizumab injections (IVR) (0.5mg/0.05ml) before vitreous surgery. IVC group means patients that received intravitreal conbercept injection (IVC) (0.5mg/0.05ml) before vitreous surgery.

SUMMARY:
Proliferative diabetic retinopathy (PDR) is the most common causes of irreversible blindness in diabetic retinopathy (DR).Although pars plana vitrectomy (PPV) is the cornerstone for treatment of advanced PDR, related postoperative complications such as recurrent VH, NVG, and postoperative fibrovascular proliferation progression may still cause serious visual impairment. Preoperative intravitreal injections of anti-VEGF drugs may represent a new strategy for making vitrectomy safer and more effective for severe PDR.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) is the most common causes of irreversible blindness in diabetic retinopathy (DR).It is characterized by progressive loss of vision, retinal edema, vitreous hemorrhage (VH), retinal neovascularization, fibrovascular proliferation, tractional retinal detachment (TRD) and neovascular glaucoma (NVG).Although pars plana vitrectomy (PPV) is the cornerstone for treatment of advanced PDR, related postoperative complications such as recurrent VH, NVG, and postoperative fibrovascular proliferation progression may still cause serious visual impairment. It is well known that vascular endothelial growth factor (VEGF) is a leading role of the neovascularization, vascular permeability, and diabetic macular edema.preoperative intravitreal injections of anti-VEGF drugs may represent a new strategy for making vitrectomy safer and more effective for severe PDR.Until now, there are two kinds of anti-VEGF drugs in China, including monoclonal antibodies, like imported drug Ranibizumab, militating by block VEGF-A, and fusion proteins, like domectic drug Conbercept, competitively inhibiting the binding of VEGF with its receptor by blocking multiple targets, VEGF-A, VEGF-B, and placental insulin-like growth factor (PlGF). Studies focusing on the comparison of efficacy between preoperative intravitreal injections of the two drugs for patients with severe PDR undergoing vitrectomy is still limited. Thus, in this study, we aim to carry out a more comprehensive comparison in intraoperative and postoperative aspects on the efficacy and safety between intravitreal ranibizumab injection (IVR) and intravitreal conbercept injection (IVC) before vitrectomy of PDR.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or more with type 1 or 2 diabetes who were clinically diagnosed with diabetic retinopathy (DR); hemoglobin A1c (HbA1c) ≤ 12%;
* persistent VH for more than 1 month or recurrent vitreous hemorrhage (VH) with or without panretinal photocoagulation (PRP);
* TRD detected by indirect ophthalmoscope or B-scan ultrasonography.

Exclusion Criteria:

* previous vitreoretinal surgeries (including vitrectomy, intravitreal drug injection) in the study eyes;
* eyes with any ocular disease that may hinder visual improvement other than PDR, such as optic atrophy or macular hole;
* history of thromboembolic events (including cerebral vascular infarctions or myocardial infarctions) or coagulation system disorders or receiving anticoagulant or antiplatelet therapy;
* eyes given gas tamponade or additional treatment like ranibizumab injection again or supplementary retinal photocoagulation during follow-up periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
BCVA | from preoperation to 3 months follow-up
  best-corrected visual acuity
CRT | from preoperation to 3 months follow-up
  central retinal thickness

SECONDARY OUTCOMES:
surgery time | during surgery
  surgery time
intraoperative bleeding | during surgery
  intraoperative bleeding
intraocular electrocoagulation use | during surgery
  intraocular electrocoagulation use
incidence of iatrogenic retinal breaks | during surgery
  incidence of iatrogenic retinal breaks
relaxing retinotomy | during surgery
  relaxing retinotomy
retinal reattachment | during surgery
  retinal reattachment
silicone oil tamponade | during surgery
  silicone oil tamponade
postoperative vitreous hemorrhage (VH) | during 3 months follow-up
  postoperative vitreous hemorrhage (VH)
neovascular glaucoma (NVG) | during 3 months follow-up
  neovascular glaucoma (NVG)
recurrent retinal detachment | during 3 months follow-up
  recurrent retinal detachment
postoperative fibrovascular proliferation progression | during 3 months follow-up
  postoperative fibrovascular proliferation progression

CONTACTS AND LOCATIONS:
Overall Officials: Jinfeng Qu, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang W, Lu J, Weng J, Jia W, Ji L, Xiao J, Shan Z, Liu J, Tian H, Ji Q, Zhu D, Ge J, Lin L, Chen L, Guo X, Zhao Z, Li Q, Zhou Z, Shan G, He J; China National Diabetes and Metabolic Disorders Study Group. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Mar 25;362(12):1090-101. doi: 10.1056/NEJMoa0908292. PMID 20335585
- [Background] Tseng VL, Greenberg PB, Scott IU, Anderson KL. Compliance with the American Academy of Ophthalmology Preferred Practice Pattern for Diabetic Retinopathy in a resident ophthalmology clinic. Retina. 2010 May;30(5):787-94. doi: 10.1097/IAE.0b013e3181cd47a2. PMID 20168268
- [Background] Bressler SB, Qin H, Melia M, Bressler NM, Beck RW, Chan CK, Grover S, Miller DG; Diabetic Retinopathy Clinical Research Network. Exploratory analysis of the effect of intravitreal ranibizumab or triamcinolone on worsening of diabetic retinopathy in a randomized clinical trial. JAMA Ophthalmol. 2013 Aug;131(8):1033-40. doi: 10.1001/jamaophthalmol.2013.4154. PMID 23807371
- [Background] Ehrlich R, Harris A, Ciulla TA, Kheradiya N, Winston DM, Wirostko B. Diabetic macular oedema: physical, physiological and molecular factors contribute to this pathological process. Acta Ophthalmol. 2010 May;88(3):279-91. doi: 10.1111/j.1755-3768.2008.01501.x. Epub 2010 Mar 11. PMID 20222885
- [Background] Wang X, Wang G, Wang Y. Intravitreous vascular endothelial growth factor and hypoxia-inducible factor 1a in patients with proliferative diabetic retinopathy. Am J Ophthalmol. 2009 Dec;148(6):883-9. doi: 10.1016/j.ajo.2009.07.007. Epub 2009 Oct 17. PMID 19837381
- [Background] Yang X, Xu J, Wang R, Mei Y, Lei H, Liu J, Zhang T, Zhao H. A Randomized Controlled Trial of Conbercept Pretreatment before Vitrectomy in Proliferative Diabetic Retinopathy. J Ophthalmol. 2016;2016:2473234. doi: 10.1155/2016/2473234. Epub 2016 Mar 13. PMID 27034822
- [Background] Cui J, Chen H, Lu H, Dong F, Wei D, Jiao Y, Charles S, Gu W, Wang L. Efficacy and Safety of Intravitreal Conbercept, Ranibizumab, and Triamcinolone on 23-Gauge Vitrectomy for Patients with Proliferative Diabetic Retinopathy. J Ophthalmol. 2018 Jun 25;2018:4927259. doi: 10.1155/2018/4927259. eCollection 2018. PMID 30046459
- [Derived] Li S, Guo L, Zhou P, Tang J, Wang Z, Zhang L, Zhao M, Qu J. Comparison of efficacy and safety of intravitreal ranibizumab and conbercept before vitrectomy in Chinese proliferative diabetic retinopathy patients: a prospective randomized controlled trial. Eye Vis (Lond). 2022 Dec 1;9(1):44. doi: 10.1186/s40662-022-00316-z. PMID 36451252